CLINICAL TRIAL: NCT00909896
Title: Prospective, Double Arm, Comparative Study for the Evaluation of Postoperative Pain, QOL, and Determination of Inflammatory Markers In Patients Undergoing Robotics Versus Open Laparotomy Approach for Staging of Endometrial Cancer
Brief Title: Study of Post Operative Pain in Endometrial Cancer Robotic Versus Laparotomy
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, David Cohn, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-08155
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Endometrial Cancer
Keywords: endometrial; pain
MeSH Terms: conditions — Endometrial Neoplasms; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Robotic Surgery candidates: Group of patients receive Robotic approach for endometrial cancer staging
- Open Laparotomy Surgical Candidates: Patients receiving open laparotomy for endometrial cancer surgical staging

SUMMARY:
This study is being done to evaluate the efficacy of robotic approach for staging of endometrial cancer as compared to an equivalent abdominal approach. The primary objective is to measure and compare postoperative pain at rest at several time points between two groups of patients undergoing either robotic or open laparotomy approach for staging of endometrial cancer.

DETAILED DESCRIPTION:
The primary objective is to measure and compare postoperative pain at rest at several time points (24 +/-4hours, 48 +/-4hours, and 72 +/-4hours) between the two groups of patients undergoing either robotic or open laparotomy approach for staging of endometrial cancer. Post operative Quality of Life will also be collected at several time points. The total amount of post operative opioid requirements during the first 24hours between patients undergoing either robotic or open laparotomy approach surgery. The survival status every four months for the first two years will be monitored, then every 6 months for up to 5 years. The primary endpoint is the mean difference in post operative pain VAS scores reported by subjects at rest at the following time points: 24+/-4, 48+/-4, and 72+/-4 hours between both groups after surgery has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects between ages 18-86 years old
* Subject provided written consent
* Preoperative diagnosis of stage i or II endometrial cancer
* Subject scheduled to undergo robotic hysterectomy or open abdominal hysterectomy at The Ohio State University
* Subject should be expected to be able to use and tolerate opioids for pain management
* Pre operative health is graded as ASA I-III
* ECOG(Eastern Cooperative Oncology Group)Performance status 0-3
* Subject willing to comply with scheduled visits

Exclusion Criteria:

* Subject is prisoner, pregnant, or under age 18 or over age 85
* Hypersensitivity to opioids
* subject is breastfeeding
* Preoperative Health grade ASA IV-V
* ECOG Performance Status 4-5
* History of receiving prior chemotherapy or radiation therapy
* Subject schedule for additional procedures at the same time as the surgical staging
* Subject with pain related illness that to the PI discretion would interfere with study assessments.
* Known history of alcohol, analgesic, or narcotic abuse within 12 months.
* Subjects taking NSAID(nonsteroidal anti inflammatory drug medications)within 7 days prior to baseline visit.
* Require and/or receive chronic analgesic therapy for any pain related condition
* Severe acute or chronic medical or psychiatric condition that would interfere with the study results.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female subjects ages 18-85 years old, Pre operative diagnosis of clinical stage I or II endometrial cancer, Subject able to tolerate use of opioids for pain management, Eastern Cooperative Oncology Group (ECOG)0-3.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2009-04-08 (Actual); Primary Completion 2013-01-29 (Actual); Study Completion 2013-01-29 (Actual)

PRIMARY OUTCOMES:
The outcome measure is mean difference in post operative pain VAS scores reported by subjects at rest at the several time points between two groups of patients undergoing either robotic or open laparotomy approach for staging of endometrial cancer. | up to 24 hours

SECONDARY OUTCOMES:
Secondary outcomes will include the measurement of post operative pain after leg extension, post operative quality of life, post operative opioid requirements during first 24hours, survival status up to five years. | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Cohn, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu